CLINICAL TRIAL: NCT06469099
Title: Ankle Injuries, Imaging and Prevention Program Effectiveness in New Army Recruits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Zinman College of Physical Education and Sports Sciences (Other)
Responsible Party: Principal Investigator, Gali Dar, Principal Investigator, University of Haifa
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 231/22
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Ankle Sprains
Keywords: soldiers; injury; ankle; exercise
MeSH Terms: conditions — Ankle Injuries; Wounds and Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: active soldiers will perform baseline examinations for the musculoskeletal system. following, an exercise intervention program will be conducted with follow-up examination at the termination of program.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- research group (Experimental): active exercises for few weeks
  Interventions: Other: excercises
- control (No Intervention): control group - no intervention, continue their routine

INTERVENTIONS:
Other: excercises — exercises for strength and balance
  Arms: research group

SUMMARY:
Infantry recruits will undergo a musculoskeletal examination to assess tendon, muscle, proprioception, agility, and joint status. Afterward, an exercise intervention program will be implemented, followed by a concluding evaluation.

DETAILED DESCRIPTION:
Purpose: To evaluate ankle injuries in new infantry recruits, including their characteristics, association with imaging and functional measures, and the effectiveness of a preventive exercise program.

Methods: 650 new male infantry soldiers aged 18-23 will be recruited to participate in the study at the beginning of their military training. At the beginning and the end of the training (after approximately six months), the soldiers will be assessed for the following: 1. Demographics (height, weight, leg length, BMI calculation), 2. Proprioception ability (Active Movement Extent Discrimination Apparatus AMEDA), 3. Dynamic balance (Y-Balance Test YBT), 4. Leg muscle strength (bilateral heel rise test), 5. Hip strength (hand-held dynamometer), 6. Ankle agility (hexagon agility hop test), 7. Ankle stability (Anterior Drawer Test, musculoskeletal ultrasound for the Anterior Talofibular Ligament), 8. Achilles tendon structure (Ultrasound tissue Characterization UTC), 9. Aerobic ability (3000 meters run, will be recorded by the fitness instructors at the training base). In addition, the soldiers will fill out a previous ankle sprains questionnaire, pre-induction physical activity questionnaire, the Cumberland Ankle Instability Tool (CAIT) for ankle perceived instability, and the Ankle Fear Avoidance Beliefs Questionnaire (ankle-FABQ).

The soldiers will perform a constructed ankle sprain prevention program for five minutes every day during the six-month length of the study. Every 1-2 weeks, the researcher will arrive at the training base to monitor ankle injuries. Those who are diagnosed with a sprain will undergo ultrasound evaluations, which will be performed every few weeks.

ELIGIBILITY:
Inclusion Criteria:

* soldiers ages 18-22

Exclusion Criteria:

* knows disease of the bones
* before orthopedic surgery

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — infantry soldiers
Enrollment: 786 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Proprioception ability | baseline, end of intervention
  Active Movement Extent Discrimination Apparatus AMEDA
balance | baseline, end of intervention
  Y balance test
Leg muscle strength | baseline, end of intervention
  bilateral heel rise test
Hip muscle strength | baseline, end of intervention
  hand held dynamometer
Ankle agility | baseline, end of intervention
  hexagon agility hop test
Ankle stability | baseline, end of intervention
  Anterior Drawer Test, musculoskeletal ultrasound for the Anterior Talofibular Ligament
Achilles tendon structure | baseline, end of intervention
  Ultrasound tissue Characterization for the percentage of fibers types

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, Prof., Principal Investigator — University of Haifa
Locations (1):
- The Academic college Levinsky-Wingate at the Wingate Institute, Netanya, Israel